CLINICAL TRIAL: NCT00091663
Title: A Multicenter, Open-Label, Phase IIIb Trial of Tarceva (Erlotinib Hydrochloride) in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate Tarceva in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: OSI3199g
Record Dates: First submitted 2004-09-15; First posted 2004-09-16 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Lung Cancer; Non-small-cell Lung Carcinoma
Keywords: Advanced non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Tarceva (erlotinib HCl)

SUMMARY:
This is a Phase IIIb, multicenter, open-label trial of daily oral Tarceva in patients with advanced (inoperable Stage IIIb or IV) NSCLC who have progressed following standard chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written (signed) informed consent(s)
* Inoperable and incurable, locally advanced, recurrent or metastatic NSCLC
* Relapse following standard chemotherapy (combination chemotherapy such as two-drug combination chemotherapy, or a single-agent chemotherapy agent for elderly or poor performance status patients)
* Age >=18 years
* ECOG performance status of 0 to 3
* Recovered from the toxic effects of prior therapy
* Able to comply with study and follow-up procedures
* Able to take oral medication
* Use of an effective means of contraception (for patients with reproductive potential)
* Granulocyte count >=1.0 x 10^9/L
* Platelet count >=75 x 10^9/L
* Serum bilirubin <1.5 x upper limit of normal (ULN)
* SGOT (AST) <2 x ULN unless elevation is clearly due to liver metastases; then SGOT (AST) must be <5 x ULN
* Serum creatinine <=1.5 mg/dL

Exclusion Criteria:

* Any unstable systemic disease (including active infection, unstable angina, congestive heart failure, myocardial infarction within the last 6 months, hepatic, renal, or metabolic disease)
* Prior therapy with any systemic HER1/EGFR small molecule inhibitor, including gefitinib (Iressa), erlotinib (Tarceva), or other investigational agents in this class
* History of another malignancy in the past 2 years unless the malignancy has been adequately treated and is associated with a 5-year anticipated survival of >=90%
* Known central nervous system (CNS) metastases that have not yet been definitively treated with surgery and/or radiation or that are symptomatic or unstable
* Nursing mothers or pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000
Dates: Start 2004-08; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (92):
- United States (92):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Hematology-Oncology Specialist, Center for Cancer Care, Huntsville, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Palo Verde Hematology/Oncology, Ltd., Glendale, Arizona
  - Arizona Hematology Oncology, PC, Tucson, Arizona
  - Little Rock Hematology Oncology Associates, Little Rock, Arkansas
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Southbay Oncology Hematology Partners, Campbell, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Cancer and Blood Institute Medical Group, Rancho Mirage, California
  - Los Palos Oncology and Hematology Center, Salinas, California
  - Naveen Gupta, MD, Inc., Upland, California
  - Hematology Oncology, PC, Stamford, Connecticut
  - Lee Cancer Clinic, Fort Myers, Florida
  - Florida Wellcare Alliance, Inverness, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Osceola Cancer Center, Kissimmee, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Mid-Florida Hematology & Oncology Centers, P.A., Orange City, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Metcare Oncology, Ormond Beach, Florida
  - Hematology Oncology Associates, Pensacola, Florida
  - Oncology and Hematology Associates of West Broward P.A., Tamarac, Florida
  - Bay Area Oncology, Tampa, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - Hematology & Oncology of NE Georgia, PC, Athens, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - Northwest Medical Specialists, Arlington Heights, Illinois
  - Hematology Oncology Consultants, Naperville, Illinois
  - Cedar Valley Medical Specialists, PC, Waterloo, Iowa
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana Oncology Associates, PMC, Lafayette, Louisiana
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - Annapolis Medical Specialists, LLC, Annapolis, Maryland
  - Maryland Hematology/Oncology Associates, PA, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, P.C., Bethesda, Maryland
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - West Michigan Regional Cancer & Blood Center, Free Soil, Michigan
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Essex Oncology of North Jersey, Belleville, New Jersey
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Combined Hematology Oncology Practice of New Jersey, Jersey City, New Jersey
  - Hematology Oncology Associates of Western Suffolk, PC, Bay Shore, New York
  - Nassau Hematology Oncology, P.C., Lake Success, New York
  - Crystal Run Healthcare, Middletown, New York
  - Westchester Hematology Oncology Associates, Mount Kisco, New York
  - Upstate NY Cancer Research and Education Foundation, Rochester, New York
  - Staten Island Medical Group, Staten Island, New York
  - Cancer Care of WNC, Asheville, North Carolina
  - Gaston Hematology and Oncology, Gastonia, North Carolina
  - Northwestern Carolina Oncology & Hematology, PA, Hickory, North Carolina
  - Piedmont Oncology Specialists, Monroe, North Carolina
  - Lake Norman Hematology/ Oncology Specialists, Mooresville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - The Gerad Center for Cancer Treatment, Lima, Ohio
  - Ohio Cancer Specialists, Inc., Mansfield, Ohio
  - Signal Point Hematology/Oncology, Inc., Middletown, Ohio
  - Comprehensive Cancer Center, Oklahoma City, Oklahoma
  - Oncology Hematology Associates of Northern Pennsylvania, PC, DuBois, Pennsylvania
  - Satish A. Shah, MD, PC, Gettysburg, Pennsylvania
  - Drs. Sambandam & Joseph Associates, Inc., Cranston, Rhode Island
  - Charleston Cancer Center, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Sioux Valley Clinic, Sioux Falls, South Dakota
  - Blue Ridge Medical Specialists, Bristol, Tennessee
  - The Family Cancer Center, Collierville, Tennessee
  - C. Michael Jones, MD PC, Germantown, Tennessee
  - McLeod Cancer & Blood Center, Johnson City, Tennessee
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Lone Star Oncology Consultants, PA, Austin, Texas
  - Coastal Bend Oncology Hematology, Corpus Christi, Texas
  - Center for Oncology Research and Treatment P. A., Dallas, Texas
  - Texas Cancer Associates, LLP, Dallas, Texas
  - Texas Hematology/Oncology Center, P.A., Dallas, Texas
  - Steve Perkins, MD, PA, Dallas, Texas
  - Utah Hematology and Oncology, Ogden, Utah
  - Rutland Regional Medical Center, Rutland, Vermont
  - Cancer Outreach Association, LLC, Abingdon, Virginia
  - Arlington Fairfax Hematology Oncology, P.C., Arlington, Virginia
  - Lynchburg Hematology Oncology Clinic, Inc., Lynchburg, Virginia
  - Cascade Cancer Center, Kirkland, Washington
  - NW Cancer Specialists, Vancouver, Washington
  - Ministry Medical Group, Rhinelander, Wisconsin

REFERENCES:
- [Result] Spigel DR, Lin M, O'Neill V, Hainsworth JD. Final survival and safety results from a multicenter, open-label, phase 3b trial of erlotinib in patients with advanced nonsmall cell lung cancer. Cancer. 2008 Jun 15;112(12):2749-55. doi: 10.1002/cncr.23490. PMID 18438878